CLINICAL TRIAL: NCT06325176
Title: Comparative Effects of Cryotherapy and Infrared Light on Pain, Redness and Healing of Episiotomy Wound
Brief Title: Comparative Effects of Cryotherapy and Infrared Light on Pain, Redness, and Healing of Episiotomy Wound
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0569
Record Dates: First submitted 2024-03-17; First posted 2024-03-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Episiotomy Wound
Keywords: cryothrapy; Episiotomy; Infrared Rays
MeSH Terms: interventions — Cryotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cryotherapy group (Experimental): During the 1st visit, the patients will be assessed for pain and episiotomy wound. The cryotherapy group will include 12 postnatal women. This group will use a bag of ice packs applied to the perineal region. The ice pack will be sealed in a plastic bag and wrapped with one layer of thin cotton tissue so that the skin of the participant will not be in direct contact with ice, which could cause discomfort. During the intervention, the women will be asked to remove their underpants and hygienic pads and remain in the dorsal recumbent position during cryotherapy that lasts 20 minutes. This procedure will be done twice a day for seven consecutive days
  Interventions: Other: Cryotherapy
- Infrared light therapy (Active Comparator): The infrared group will include 12 postnatal women they will be encouraged to place an infrared lamp at a distance of 45 cm from the perineum and the heat produced with 230 volts for twenty minutes. But the mother is checked after the first five minutes to make sure that she is not being burned. The researcher will demonstrate for each woman how to use an infrared lamp, and it will be followed by re-demonstrations and discussions. These procedures will be carried out in the morning and evening for seven consecutive days. The researcher gives the infrared lamp device to each woman and then restores it after completion of the study
  Interventions: Device: Infrared light therapy

INTERVENTIONS:
Other: Cryotherapy — During the 1st visit of the patients, they will be assessed for pain and episiotomy wound. The cryotherapy group will include 12 postnatal women. This group will use a bag of ice pack applied to the perineal region. The ice pack will be sealed in plastic bag and wrapped with one layer of a thin cotton tissue so that the skin of the participant would not be in direct contact with ice, which could cause discomfort. During the intervention, the women will be asked to remove their underpants and hygienic pads and remain in the dorsal recumbent position during cryotherapy that lasted 20 minutes. This procedure will be done twice a day for seven consecutive days
  Arms: Cryotherapy group
Device: Infrared light therapy — Infrared group will include 12 postnatal women they will encourage to place an infrared lamp at distance of 45 cm from the perineum and the heat produced with 230 volts for twenty minutes. But the mother is checked after the first five minutes to make sure that she was not being burned. The researcher will demonstrate for each woman how to use infrared lamp, and it will be followed by re demonstrations and discussions. These procedures will carry out in the morning and evening for seven consecutive days. The researcher gives the infrared lamp device for each woman then restore it after completion of the study
  Arms: Infrared light therapy

SUMMARY:
The study will be a randomized clinical trial and will be conducted in Bahawalpur Victoria Hospital, Bahawalpur. The subjects (n=24) will be divided into two groups. Group A will include 12 postnatal women and for treatment, cryotherapy will be applied for 20 minutes. Group B will include 12 women and receive infrared light, an infrared lamp will be put at a distance of 45 cm from the perineum, and the heat produced with 230 volts for twenty minutes. The participant will be checked after the first five minutes to make sure that she is not being burned. This procedure will be done twice a day for 7 consecutive days.

DETAILED DESCRIPTION:
One of the most often used delivery methods is the episiotomy. Severe side effects like infection, dehiscence of the incision, and perineal discomfort are possible. In addition to increased blood loss during birth, mothers who undergo episiotomy have the risk of experiencing delayed wound healing along with increased pain in the early puerperium. After birth, episiotomy treatment begins right away and would involve both pain management and local wound care. The data will be assessed on the baseline 3rd day and 7th day of treatment. A numeric pain rating scale (NPRS) will be used to assess the severity of Pain. REEDA scale will be used for Redness, Edema, Ecchymosis, Discharge, and Approximation (closeness of skin edges). SPSS version 25 will be used for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Women who underwent episiotomy between 6 to 24 hours postpartum.
* Delivered a live baby.
* Complete full-term labor.
* episiotomy type medial and Medio-lateral.
* primiparous women and multiparous women.

Exclusion Criteria:

Used pain-relieving drugs.

* Women with diabetes and pre-eclampsia.
* Febrile conditions.
* Severe infection.
* Chronic medical conditions that may affect wound healing.
* Allergies and sensitivity to heat/cold.
* Recent surgery of pelvis or abdomen.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 24 (Actual)
Dates: Start 2024-03-20 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | up to 1 week
  The NPRS is a segmented numeric scale in which the respondent selects a whole number(0-10 integers) that best reflects the intensity of his/her pain. The common format is a horizontal bar or line. NPRS is anchored by terms describing pain severity extremes.
The standardized REEDA scale: | up to 1 week
  The REEDA scale is an observational check list used for assessing perineal healing.The acronym REEDA is derived from five components: Redness, Edema, Ecchymosis, Discharge and Approximation of the wound edges.Each component takes a score ranged from 0 to 3. Higher score indicates poor wound healing while lower score indicates good wound healing.The total score of REEDA scale was categorized as follows:
  0 to 2 - Healed.3 to 5 - Moderately healed.6 to 8- Mildly healed.9 to 15 - Not healed.

CONTACTS AND LOCATIONS:
Overall Officials: Mutieba Javed, MS*, Principal Investigator — Riphah International University, Lahore, Pakistan
Locations (1):
- Bahawalpur Victoria Hospital(BVH), Chak Four Hundred Fifty-four, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zakariaee SS, Shahoei R, Hashemi Nosab L, Moradi G, Farshbaf M. The Effects of Transcutaneous Electrical Nerve Stimulation on Post-Episiotomy Pain Severity in Primiparous Women: A Randomized, Controlled, Placebo Clinical Trial. Galen Med J. 2019 Aug 14;8:e1404. doi: 10.31661/gmj.v8i0.1404. eCollection 2019. PMID 34466506
- [Background] Choudhari RG, Tayade SA, Venurkar SV, Deshpande VP. A Review of Episiotomy and Modalities for Relief of Episiotomy Pain. Cureus. 2022 Nov 17;14(11):e31620. doi: 10.7759/cureus.31620. eCollection 2022 Nov. PMID 36540434
- [Background] Solt Kirca A, Korkut Oksuz S, Murat N. The effect of cold application on episiotomy pain: A systematic review and meta-analysis. J Clin Nurs. 2022 Mar;31(5-6):559-568. doi: 10.1111/jocn.15912. Epub 2021 Jun 13. PMID 34121251
- [Background] Roma NZH, Essa RM, Rashwan ZI, Ahmed AH. Effect of Dry Heat Application on Perineal Pain and Episiotomy Wound Healing among Primipara Women. Obstet Gynecol Int. 2023 Jan 4;2023:9572354. doi: 10.1155/2023/9572354. eCollection 2023. PMID 36643188
- [Background] Beleza ACS, Ferreira CHJ, Driusso P, Dos Santos CB, Nakano AMS. Effect of cryotherapy on relief of perineal pain after vaginal childbirth with episiotomy: a randomized and controlled clinical trial. Physiotherapy. 2017 Dec;103(4):453-458. doi: 10.1016/j.physio.2016.03.003. Epub 2016 Nov 9. PMID 27956033